CLINICAL TRIAL: NCT00004930
Title: Phase I and Clinical Pharmacologic Study of Inhaled Doxorubicin in Adults With Advanced Solid Tumors Affecting the Lungs
Brief Title: Inhaled Doxorubicin in Treating Patients With Primary Lung Cancer or Lung Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-049; CDR0000067614 (Registry Identifier: PDQ (Physician Data Query)); BMI-98-DOX-001; NCI-G00-1696
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: recurrent non-small cell lung cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; lung metastases; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Doxorubicin

INTERVENTIONS:
Drug: doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of inhaled doxorubicin in treating patients who have primary lung cancer or lung metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and phase II dose of inhaled doxorubicin administered every 3 weeks in patients with primary lung cancer or cancer metastatic to the lung.
* Determine the toxic effects and pharmacokinetic profile of this regimen in this patient population.
* Examine the relationship between pharmacodynamic parameters and toxic effects of this regimen in these patients.
* Obtain preliminary evidence of therapeutic activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive inhaled doxorubicin every 3 weeks. Treatment continues for a maximum of 3 courses in the absence of unacceptable toxicity or disease progression. Patients may reenter at a higher dose level after a 3-month waiting period.

Cohorts of 3-6 patients receive escalating doses of doxorubicin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 6 weeks.

PROJECTED ACCRUAL: A total of 3-36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary lung cancer or cancer metastatic to the lung that is not potentially curable by standard chemotherapy, radiotherapy, or surgery

  * Bronchoalveolar cell lung cancer allowed
* Lung metastases from soft tissue sarcoma allowed
* No leukemia or lymphoma

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 160,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin no greater than 1.0 mg/dL
* AST/ALT less than 1.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.2 mg/dL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* LVEF normal by MUGA scan or echocardiography
* No unstable angina
* No congestive heart failure
* No symptomatic arrhythmias

Pulmonary:

* DLCO at least 65% of normal
* FVC at least 50% predicted
* FEV1 at least 50% predicted
* Resting oxygen saturation at least 90%
* Exercise oxygen saturation at least 85%
* No complete atelectasis
* No asthma

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study
* No congenital problems (e.g., cleft palate) or other anomalies that would prevent tight fit of mouth seal
* No other concurrent illness that would preclude study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy and recovered
* No prior bleomycin or nitrosoureas
* No prior mitomycin greater than 25 mg/m^2
* No prior anthracyclines greater than 450 mg/m^2
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* No prior chest (pulmonary or mediastinal) or thoracic spine radiotherapy

  * Patients with only chest wall or primary breast radiation are eligible
* No concurrent thoracic irradiation

Surgery:

* See Disease Characteristics
* No prior pneumonectomy

Other:

* No daily or as necessary respiratory drugs via inhaler or nebulizer
* No other concurrent experimental drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-07; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naiyer Rizvi, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio